CLINICAL TRIAL: NCT03471156
Title: Persistent Pain After Colonic Endoscopic Mucosal Resection: Predictors, a Management Algorithm and Outcomes
Brief Title: Prospective Evaluation of Pain Assessment and Management Protocol for Post-procedural Pain After Endoscopic Mucosal Resection of Colonic Polyps >20mm
Status: Completed | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Clinical Professor of Medicine, Western Sydney Local Health District
Other Study IDs: LNR/15/WMEAD/25
Record Dates: First submitted 2017-07-09; First posted 2018-03-20 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Pain; Endoscopic Mucosal Resection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post EMR: Patients are observed post EMR procedure for pain. Standard of care data is collected

SUMMARY:
Endoscopic mucosal resection (EMR) of large (≥20 mm) laterally spreading colonic lesions (LSL) is safe, effective and superior to surgery. This advantage is based on a day stay model of care, however the most common adverse event is abdominal pain and this is a major impediment to this efficiency. No prospective data exist on the optimal selection of analgesics, the necessary recovery period or the triggers that should alert the practitioner to a more serious trajectory and the need for escalation of care.

We aimed to characterise potential predictors for persistent (>5 minutes) post-procedural pain (PP) and develop a simple and effective management algorithm for patients with PP based on the need for analgesics in recovery.

Data on consecutive patients with a LSL referred for EMR at a single, tertiary referral centre were included. Patient and lesion characteristics and peri-procedural data were prospectively collected. Standard post EMR care included 2 hours in first stage recovery followed by 1 hour in 2nd stage recovery where clear fluids were given and discharge after if the patients were well. PP was graded from 0 to 10 using a Visual Analogue Scale (VAS). If PP occurred >5 minutes, 1 gram of paracetamol was administered parenterally and outcomes were monitored. If pain settled the patient was transferred to second stage recovery after medical review. PP >30 minutes lead to clinical review and upgrade of analgesics to fentanyl, with a starting dose of 25 micrograms (mcg) up to a maximum of 100 mcg. Investigations, admission and interventions for PP are recorded.

DETAILED DESCRIPTION:
Large, sessile, colonic polyps of ≥ 20 mm are at increased risk of progressing to colorectal cancer (CRC). Most colonic polyps are small and pedunculated and can be safely removed by conventional polypectomy. Treatment of large polyps however, is challenging but very important in preventing development of CRC, the second leading cause of cancer deaths worldwide. Early detection and treatment of these polyps, possible through vigilant CRC screening via colonoscopy, shows significant reduction in incidence of CRC.

Over the last decade, endoscopic mucosal resection (EMR) has been recognised as a safe and reliable alternative to surgery to remove large, sessile colonic polyps of ≥ 20mm. The benefits of EMR over traditional surgery include reduced risk of peri- and post-operative complications from surgery (particularly in elderly patients with multiple co-morbidities), less health expenditure and reduced length of hospital admission. The majority of patients can be managed safely as outpatients post EMR.

EMR has been proven to be a safer alternative to traditional surgery, but is a technically challenging procedure. The most common complication post procedure is non-specific abdominal pain, which occurs in 10-20% of cases. The cause is often innocent such as simple luminal distension during the procedure. The advent of improved EMR techniques, for example using carbon dioxide instead of air insufflation, significantly reduces incidence of abdominal pain and subsequently need for admission.

Colonic perforation during colonoscopy rates range from 0.06 to 0.1%. Advanced age, female gender, having a colonoscopy indication of abdominal pain or Crohn's disease, result in a statistically higher risk of colonic perforation. In addition, ICU inpatients have substantially greater odds of perforation. A recent study, conducted over twelve years in a total of 110,785 patients undergoing diagnostic and therapeutic colonoscopies, showed one case of colonic perforation associated with EMR.

Currently, it remains difficult to delineate innocent abdominal pain from more serious complications. There are no standard algorithms used in clinical practice to stratify risk post EMR according to patient's symptoms and there are no data supporting previously proposed pain algorithms. There is also a paucity of data regarding pain scales employed in the past to show significant correlation between pain level and risk of perforation or bleeding. The 100mm Visual Analog Scale (VAS) has been documented to have sound correlation in patients presenting to the emergency department with an acute abdomen and could be a useful aid in a formal assessment based on pain post EMR.

With the prospectively recorded data in this study, we aim to validate an algorithm to provide decision support in first stage recovery of Endoscopy Departments. This algorithm on assessment and management of post EMR pain, will identify patients at risk for more serious complications, and will allow health carers to recognize these complications and act more accurately. Ultimately, this will improve patient's outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to Westmead Hospital Endoscopy Unit to undergo an EMR of a colonic lesion reported to be ≥20mm in size.
* Age ≥18 years.
* Patients able to give informed consent to involvement in the trial. For patients who do not speak English, an interpreter will be asked to translate the informed consent.

Exclusion Criteria:

Inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data on consecutive patients with a LSL referred for EMR at a single, tertiary referral centre were included. Patient and lesion characteristics and peri-procedural data were prospectively collected. Standard post EMR care included 2 hours in first stage recovery followed by 1 hour in 2nd stage recovery where clear fluids were given and discharge after if the patients were well. PP was graded from 0 to 10 using a Visual Analogue Scale (VAS). If PP occurred >5 minutes, 1 gram of paracetamol was administered parenterally and outcomes were monitored. If pain settled the patient was transferred to second stage recovery after medical review. PP >30 minutes lead to clinical review and upgrade of analgesics to fentanyl, with a starting dose of 25 micrograms (mcg) up to a maximum of 100 mcg. Investigations, admission and interventions for PP were recorded.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with EMR related pain post-procedurally | up to 24 hours
  Patients are observed for pain post-procedurally and data collected on when/how pain is relieved

SECONDARY OUTCOMES:
Correlate post-procedural pain with procedural data | up to 24 hours
  Identify if any patient or lesion factors are predictive of post EMR pain

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Desomer L, Tate DJ, Pillay L, Awadie H, Sidhu M, Ahlenstiel G, Bourke MJ. Intravenous paracetamol for persistent pain after endoscopic mucosal resection discriminates patients at risk of adverse events and those who can be safely discharged. Endoscopy. 2023 Jul;55(7):611-619. doi: 10.1055/a-2022-6530. Epub 2023 Jan 30. PMID 36716781